CLINICAL TRIAL: NCT03470987
Title: The Role of Visfatin Levels in Gingival Crevicular Fluid as Potential Biomarker in The Relationship Between Obesity and Periodontal Disease
Brief Title: The Role of Visfatin in Obesity and Periodontal Disease
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Deniz Cetiner, Principal Investigator, Gazi University
Other Study IDs: OBESITY
Record Dates: First submitted 2018-03-06; First posted 2018-03-20 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Periodontitis
Keywords: obesity; periodontitis; cytokines
MeSH Terms: conditions — Obesity; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gingival crevicular fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1:nO-Ctrl: Non-obese patients without generalized chronic periodontitis who were undergone Phase I periodontal therapy
  Interventions: Procedure: Phase I Periodontal therapy
- Group 2:nO-CP: Non-obese patients with generalized chronic periodontitis who were undergone Phase I periodontal therapy
  Interventions: Procedure: Phase I Periodontal therapy
- Group 3: O-Ctrl: Obese patients without generalized chronic periodontitis who were undergone metabolic control and Phase I periodontal therapy
  Interventions: Procedure: Phase I Periodontal therapy; Dietary Supplement: Metabolic control
- Group 4: O-CP: Obese patients with generalized chronic periodontitis who were undergone metbolic control and Phase I periodontal therapy
  Interventions: Procedure: Phase I Periodontal therapy; Dietary Supplement: Metabolic control

INTERVENTIONS:
Procedure: Phase I Periodontal therapy — Oral hygiene instuction, scaling and root planning
Dietary Supplement: Metabolic control — Calorie restricted diet
  Groups: Group 3: O-Ctrl; Group 4: O-CP

SUMMARY:
Visfatin is an adipokine that plays an important role in immune functions as a growth factor, enzyme, and proinflammatory mediator. The investigators aimed to determine the levels of visfatin, interleukin-6 (IL-6) and tumor necrosis factor-alpha (TNF-alpha) in gingival crevicular fluid (GCF) in both obese/non-obese patients, with/without generalized chronic periodontitis (GCP). Patients were categorized as obese (O) (n=31) or non-obese (nO) (n=19). Groups were divided into four subgroups according to periodontal conditions: (1) periodontally healthy without obesity (nO-Ctrl); (2) GCP without obesity (nO-CP); (3) periodontally healthy with obesity (O-Ctrl); and (4) GCP with obesity (O-CP). Demographic variables and anthropometric and laboratory data were recorded. Periodontal measurements were recorded at baseline and 3rd months after either non-surgical periodontal treatment or calorie restricted diet therapy. At the same time GCF samples were taken from patients to analyze TNF-alpha, IL-6, and visfatin levels.

DETAILED DESCRIPTION:
Overweightness and obesity are defined as the accumulation of fat in body tissues that might impair overall health. Adults are considered overweight if their body mass index (BMI, calculated as weight in kg/[height in meters]2) is ≥ 25 and obese if BMI ≥ 30 kg/m2. The prevalence of overweightness and obesity has increased worldwide during recent decades.

Obesity is usually related to a chronic low-grade systemic inflammation resulting in significant changes in the concentrations of cytokines and hormones, which subsequently leads to the development of obesity-linked disorders, including insulin resistance, type II diabetes, cardiovascular diseases, dyslipidemia, and metabolic syndrome. Since the host response is among the most crucial factors affecting the pathogenesis of periodontal disease, multiple studies have addressed the possible associations between BMI, overweightness, obesity, diabetes, the serum level of lipids, cholesterol, and periodontal breakdown, with mixed results. Many studies have demonstrated a positive association between obesity and periodontitis and suggested that obesity-related inflammation might promote periodontitis by secretion of inflammatory markers by the adipose tissue, which might subsequently increase gingival inflammation. The association between obesity and periodontal disease is based on the amassing of white adipose tissue (WAT) and increased secretion levels of adipokines from WAT.

WAT is an energy storage organ with some metabolic activities, participating in the endocrine and secretory systems. WAT secretes several immune-modulatory adipokine molecules, such as adiponectin, leptin, visfatin, resistin, chemerin, tumor necrosis factor-alpha (TNF-alpha), interleukin-1β (IL-1β), and interleukin-6 (IL-6). It has been found that these molecules are involved in a wide range of physiologic and pathologic processes, including immunity and inflammation. Thus, cytokines and hormones released from adipose tissue might play a role in the destruction of periodontal tissue by inducing hyperinflammatory responses.

Visfatin is a multi-potential mediator that functions as a growth factor, cytokine, an enzyme with a role in energy metabolism, and as a proinflammatory mediator. It is mainly released from adipose tissue, especially from macrophages, and can also be released from lymphocytes, dendritic, muscle, and bone marrow cells. Visfatin has an important role in the regulation of the immune response. Visfatin inhibits neutrophil apoptosis during inflammation and increases TNF-alpha, IL-1β, and IL-6 levels. The expression of visfatin is increased under inflammatory conditions, such as rheumatoid arthritis, cardiovascular diseases, type-II diabetes mellitus, and periodontal disease.

Although several studies have demonstrated the relationship between periodontitis and obesity, no study has evaluated the levels of visfatin in gingival crevicular fluid (GCF) in obese individuals with periodontitis. Increased adipocytes levels, such as visfatin, cause secretion of cytokines, which are known to play an important role in periodontitis, and might trigger periodontitis formation and development.

Therefore, the main objective of this study was to analyze the levels of visfatin, IL-6, and TNF-alpha in obese and non-obese individuals, with or without generalized chronic periodontitis (GCP). Secondarily, the investigators aimed to evaluate metabolic and clinical periodontal parameters, and also clarify the relationship between these parameters and adipocytokines. The hypothesis is that adipocytokine molecules are involved in the pathogenesis of inflammatory diseases; if true, individuals who are obese with periodontitis would present increased levels of visfatin, IL-6, and TNF-alpha in their GCF.

ELIGIBILITY:
Inclusion Criteria:

* having > 22 natural teeth
* no systemic diseases
* having good cooperation
* having BMI > 30
* waist circumference > 88 cm for females for obese patients
* waist circumference > 102 cm for males for obese patients
* age > 20 years

Exclusion Criteria:

* presence of localized chronic periodontitis
* received periodontal therapy/surgery in the previous 6 months
* pregnancy
* use of any hormone therapy
* history of antibiotic or anti-inflammatory drugs therapy within the previous 6 months
* current and former smoker
* lactation
* presence of aggressive periodontitis
* presence of periapical pathologies

Ages: 20 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The 195 patients diagnosed with obesity in the outpatient clinics of Endocrinology and Metabolic Diseases Department, Ataturk Hospital, Turkey, were potential candidates and were interviewed according to our case definition and invited to be included in the study. Thirty-one of 195 volunteers accepted and signed the informed study protocol and took part in the study. All individuals were thoroughly informed of the nature, potential risks, and benefits of their participation in the study before providing their informed consent.
  In the same period, 100 consecutive non-obese patients were screened from the Department of Periodontology, Faculty of Dentistry, Gazi University, Turkey, who were systemically healthy and fulfilled the inclusion criteria, of which 19 agreed to participate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Cytokine levels in Gingival crevicular fluid | Beginning of the study (baseline) and 3 months following Phase I periodontal therapy and metbolic control
  Gingival crevicular fluid samples were collected at baseline and repeated at 3rd months following Phase I periodontal therapy and metabolic control.
  In the periodontally healthy group, samples were obtained from maxillary anterior four teeth exhibiting probing depth < 3mm without clinical attachment level or bleeding on probing. Four sites from each tooth were used for Gingival crevicular fluid sampling.
  In the generalized chronic periodontitis groups, Gingival crevicular fluid samples were collected from four teeth with bleeding on probing, probing depth≥ 5 mm, clinical attachment level≥ 5 mm, and 30% bone loss. Visfatin, TNF alpha and IL-6 levels in these fluid samples were determined using an enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Clinical attachment level | Change from baseline clinical attachment level to 3rd month level
  Clinical attachment level which is the position of the soft tissue in relation to the cemento-enamel junction was noted from all teeth, excluding third molars at the baseline and 3 months following Phase I periodontal therapy and metabolic control
Probing depth | Change from baseline probing depth value at 3rd month value
  Probing depth was noted from all teeth, excluding third molars, on midbuccal and midlingual sites and the buccal aspects of the interproximal contact area for mesial and distal sites using a William's periodontal probe at baseline and 3 months following Phase I periodontal therapy and metabolic control
Bleeding on probing | Change from baseline bleeding on probing score to 3rd month score
  The presence of bleeding after probing was noted from all teeth, excluding third molars at the baseline and 3 months following Phase I periodontal therapy and metabolic control
Gingival index | Change from baseline gingival index score to 3rd month score
  The gingival index which is a measure of periodontal disease based on the severity and location of the lesion was noted from all teeth, excluding third molars at the baseline and 3 months following Phase I periodontal therapy and metabolic control
Plaque index | Change from baseline plaque index score to 3rd month score
  The plaque index which is an index for estimating the status of oral hygiene by measuring dental plaque that occurs in the areas adjacent to the gingival margin was noted from all teeth, excluding third molars at the baseline and 3 months following Phase I periodontal therapy and metabolic control

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Cetiner, Prof, Study Chair — Gazi University Faculty of Dentistry Department of Periodontology
Locations (1):
- Gazi University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keller A, Rohde JF, Raymond K, Heitmann BL. Association between periodontal disease and overweight and obesity: a systematic review. J Periodontol. 2015 Jun;86(6):766-76. doi: 10.1902/jop.2015.140589. Epub 2015 Feb 12. PMID 25672656
- [Background] Suvan J, D'Aiuto F, Moles DR, Petrie A, Donos N. Association between overweight/obesity and periodontitis in adults. A systematic review. Obes Rev. 2011 May;12(5):e381-404. doi: 10.1111/j.1467-789X.2010.00808.x. Epub 2011 Feb 23. PMID 21348914
- [Background] Al-Zahrani MS, Bissada NF, Borawskit EA. Obesity and periodontal disease in young, middle-aged, and older adults. J Periodontol. 2003 May;74(5):610-5. doi: 10.1902/jop.2003.74.5.610. PMID 12816292
- [Background] Goncalves TE, Zimmermann GS, Figueiredo LC, Souza Mde C, da Cruz DF, Bastos MF, da Silva HD, Duarte PM. Local and serum levels of adipokines in patients with obesity after periodontal therapy: one-year follow-up. J Clin Periodontol. 2015 May;42(5):431-9. doi: 10.1111/jcpe.12396. Epub 2015 Apr 30. PMID 25858047
- [Background] Zimmermann GS, Bastos MF, Dias Goncalves TE, Chambrone L, Duarte PM. Local and circulating levels of adipocytokines in obese and normal weight individuals with chronic periodontitis. J Periodontol. 2013 May;84(5):624-33. doi: 10.1902/jop.2012.120254. Epub 2012 Jul 27. PMID 22839694
- [Background] Trayhurn P, Beattie JH. Physiological role of adipose tissue: white adipose tissue as an endocrine and secretory organ. Proc Nutr Soc. 2001 Aug;60(3):329-39. doi: 10.1079/pns200194. PMID 11681807
- [Background] Balli U, Ongoz Dede F, Bozkurt Dogan S, Gulsoy Z, Sertoglu E. Chemerin and interleukin-6 levels in obese individuals following periodontal treatment. Oral Dis. 2016 Oct;22(7):673-80. doi: 10.1111/odi.12520. Epub 2016 Jul 11. PMID 27265537
- [Background] Vazquez-Vela ME, Torres N, Tovar AR. White adipose tissue as endocrine organ and its role in obesity. Arch Med Res. 2008 Nov;39(8):715-28. doi: 10.1016/j.arcmed.2008.09.005. PMID 18996284
- [Background] Wozniak SE, Gee LL, Wachtel MS, Frezza EE. Adipose tissue: the new endocrine organ? A review article. Dig Dis Sci. 2009 Sep;54(9):1847-56. doi: 10.1007/s10620-008-0585-3. Epub 2008 Dec 4. PMID 19052866
- [Background] Kloting N, Bluher M. Adipocyte dysfunction, inflammation and metabolic syndrome. Rev Endocr Metab Disord. 2014 Dec;15(4):277-87. doi: 10.1007/s11154-014-9301-0. PMID 25344447
- [Background] Costford SR, Bajpeyi S, Pasarica M, Albarado DC, Thomas SC, Xie H, Church TS, Jubrias SA, Conley KE, Smith SR. Skeletal muscle NAMPT is induced by exercise in humans. Am J Physiol Endocrinol Metab. 2010 Jan;298(1):E117-26. doi: 10.1152/ajpendo.00318.2009. Epub 2009 Nov 3. PMID 19887595
- [Background] Ritchie CS. Obesity and periodontal disease. Periodontol 2000. 2007;44:154-63. doi: 10.1111/j.1600-0757.2007.00207.x. No abstract available. PMID 17474931